CLINICAL TRIAL: NCT00180258
Title: Comparison of Medical Therapy, Pacing and Defibrillation in Heart Failure
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Clinicals0002
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2007-01-25 (Estimated); Status verified 2007-01

CONDITIONS: Congestive Heart Failure
Keywords: Cardiac Resynchronization Therapy (CRT); Heart Failure; Defibrillator; Pacemaker
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy; Defibrillators

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy with & without defibrillator

SUMMARY:
The purpose of this study is to determine whether combined mortality and hospitalization in heart failure patients receiving optimal pharmacologic therapy can be reduced by combining optimal pharmacologic therapy and 1) biventricular pacing therapy alone or 2) biventricular pacing with defibrillation.

DETAILED DESCRIPTION:
Evaluation of new therapies for the treatment of heart failure should address mortality, morbidity, hospitalization, and cardiac symptoms and function when compared to standard pharmacologic therapy. The COMPANION trial is designed to address all of these objectives. This clinical investigation is an open-label, prospective, multi-center, randomized clinical trial. Every patient enrolled in the study is to be prescribed to optimal pharmacologic heart failure therapy, as tolerated, regardless of randomization.

ELIGIBILITY:
Inclusion Criteria:

* Moderate or severe heart failure, defined as symptomatic heart failure for at least six months with NYHA Class III or IV symptoms at the time of enrollment, AND at least one of the following events in the previous 12 months:
* Hospitalization for heart failure management
* Outpatient visit in which intravenous (IV) inotropes or vasoactive infusion were administered continuously for at least 4 hours
* Emergency room visit of at least twelve hours duration in which IV heart failure medications were administered (including diuretics)
* QRS > or = 120 ms and PR interval > 150 ms from any two leads of a 12-lead ECG
* Left ventricular ejection fraction < or = 35%
* Left ventricular end diastolic dimension > or = 60 mm (required only if LVEF measured by echo) or > 3.0 cm/m2 [The cm/m2 is calculated by LVEDD (in cm) divided by BSA (body surface area)].
* Age > or = 18 years
* Optimal pharmacologic therapy for heart failure

Exclusion Criteria:

* Unable or unwilling to undergo device implant and follow-up testing
* Meet the general indications for an implantable cardioverter defibrillator
* Meet the general indications for antibradycardia pacing
* Expected to receive a heart transplant in the next six months
* Chronic, medically refractory atrial tachyarrhythmias
* Unexplained syncope
* Myocardial infarction within 60 days of randomization
* History of non-compliance with oral heart failure therapy
* Progressive or unstable angina
* Uncontrolled blood pressure: Systolic BP > 160 mm Hg or < 85 mm Hg or diastolic BP > 90 mm Hg
* Patients with a hypersensitivity to a 0.7 mg nominal dose of dexamethasone acetate
* Surgically uncorrected primary valvular heart disease
* Coronary artery disease (CAD) in which surgical or percutaneous correction is recent (within 60 days of randomization)
* Women who are pregnant or not using medically acceptable birth control
* Hypertrophic obstructive cardiomyopathy
* Amyloid disease
* Hospitalization for heart failure or IV inotropic or vasoactive therapy in excess of 4 hours in the 30 days prior to enrollment
* Have a tricuspid prosthesis
* Involved in any other investigational studies
* Life expectancy < 6 months due to any other medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2200
Dates: Start 2000-01; Study Completion 2002-12

PRIMARY OUTCOMES:
Combination of all-cause mortality and first hospitalization (time to first event), where all-cause mortality is defined as death from all causes.

SECONDARY OUTCOMES:
Total survival for both the CONTAK CD and CONTAK TR CHFDs when used in conjunction with pharmacologic therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple locations in the US, Saint Paul, Minnesota, United States

REFERENCES:
- [Result] Bristow MR, Saxon LA, Boehmer J, Krueger S, Kass DA, De Marco T, Carson P, DiCarlo L, DeMets D, White BG, DeVries DW, Feldman AM; Comparison of Medical Therapy, Pacing, and Defibrillation in Heart Failure (COMPANION) Investigators. Cardiac-resynchronization therapy with or without an implantable defibrillator in advanced chronic heart failure. N Engl J Med. 2004 May 20;350(21):2140-50. doi: 10.1056/NEJMoa032423. PMID 15152059
- [Derived] Cleland JGF, Bristow MR, Freemantle N, Olshansky B, Gras D, Saxon L, Tavazzi L, Boehmer J, Ghio S, Feldman AM, Daubert JC, de Mets D. The effect of cardiac resynchronization without a defibrillator on morbidity and mortality: an individual patient data meta-analysis of COMPANION and CARE-HF. Eur J Heart Fail. 2022 Jun;24(6):1080-1090. doi: 10.1002/ejhf.2524. Epub 2022 May 22. PMID 35490339
- [Derived] Anand IS, Carson P, Galle E, Song R, Boehmer J, Ghali JK, Jaski B, Lindenfeld J, O'Connor C, Steinberg JS, Leigh J, Yong P, Kosorok MR, Feldman AM, DeMets D, Bristow MR. Cardiac resynchronization therapy reduces the risk of hospitalizations in patients with advanced heart failure: results from the Comparison of Medical Therapy, Pacing and Defibrillation in Heart Failure (COMPANION) trial. Circulation. 2009 Feb 24;119(7):969-77. doi: 10.1161/CIRCULATIONAHA.108.793273. Epub 2009 Feb 9. PMID 19204305